CLINICAL TRIAL: NCT02077309
Title: Linagliptin as a Modulator of Vascular Inflammation in Patients With Type 2 Diabetes Mellitus
Brief Title: Effect of Linagliptin on Vascular Inflammation in Patients With Type 2 Diabetes Mellitus
Acronym: Lina-Plaque
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: bad recruitment of suitable participants, just 4 patients in one year
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-027; 111/13 (Other: Ethic Commitee); 2012-003859-12 (EudraCT Number)
Record Dates: First submitted 2014-02-28; First posted 2014-03-04 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2015-12

CONDITIONS: Diabetes Mellitus Type 2 (T2DM); Vascular Inflammation; Plaque Morphology
Keywords: T2DM,; vascular inflammation,; 18-FDG-PET,; plaque morphology,; MRI,; DPP-4 Inhibition
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Linagliptin (Active Comparator): Patients will receive 5 mg linagliptin once daily for a period of 6 months.
  Interventions: Drug: Linagliptin
- Placebo (Placebo Comparator): Patients will take placebo tablets once daily for a period of 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Linagliptin
  Other Names: Trade name Trajenta® by Boehringer Ingelheim (BI) Pharma GmbH & Co KG, Biberach, Germany
  Arms: Linagliptin
Drug: Placebo
  Other Names: Produced by Boehringer Ingelheim (BI) Pharma GmbH & Co KG, Biberach, Germany
  Arms: Placebo

SUMMARY:
Examination of the effect of Linagliptin versus placebo for 6 months on vascular inflammation of the carotic artery and on abdominal adipose tissue inflammation in patients with diabetes mellitus type 2. The effect will be assessed by FDG-PET scan.

Furthermore the effect of Linagliptin on the vessel wall volume of the carotid artery will be assessed by MRI scan and biomarkers of vascular inflammation will be analyzed in blood samples.

DETAILED DESCRIPTION:
As part of the screening a PET-CT scan is executed to examine baseline vascular inflammation of the carotid artery and to evaluate abdominal adipose tissues inflammation.

Patients who are eligible to participate in the study according to the in- and exclusion criteria will be randomised in one of the two study arms.

According to the randomisation the patients will receive 5 mg Linagliptin or placebo per day for a period of 6 months.

To evaluate the effect of Linagliptin versus placebo the vessel wall volume of the artery will be assessed by MRI scan and the vascular inflammation of the carotid artery by FDG-PET, furthermore the vascular inflammation will be analyzed by biomarkers in blood samples and the abdominal adipose tissue inflammation will investigated by subcutaneous adipose tissue biopsies.

ELIGIBILITY:
Inclusion Criteria:

1. Diabetes mellitus Type 2
2. HbA1c > 7%
3. Age > 50 years
4. Coronary artery disease or carotid artery disease
5. 18F-FDG uptake of the carotid arterial wall to background (blood) ratio > 1.8
6. Written informed consent prior to study participation
7. Stable anti-diabetic and cholesterol lowering medication for the last 3 month
8. Stable anti-diabetic medication for the last 6 weeks which should include a maximal tolerated dose of metformin (unless contraindication or intolerance to metformin does exist);
9. Indication to increase anti-diabetic medication as judged by the investigator

Exclusion Criteria:

1. Diabetes mellitus type 1
2. Use of DPP-4 Inhibitor, GLP-1 agonists, Thiazolindinedione
3. Kidney disease CKD 4 and more (GFR < 30 ml/min/1.73)
4. Liver disease (ALT or AST > 3 times the upper limit of norm) or known liver cirrhosis
5. Any reason for not being able to sustain the imaging studies
6. Pacemaker/ICD/metallic clips in close relation to vessels in the brain
7. Uncontrolled thyroid disease
8. Active malignant disease
9. Chronic inflammatory disease
10. Chronic use of NSAR or cortison
11. HbA1c > 8.5%
12. Recent (<3 months) clinically significant coronary or cerebral vascular event
13. Pregnant females as determined by positive [serum or urine] HCG test at Screening or prior to dosing
14. Lactating females
15. The subject has a history of any other illness, which, in the opinion of the Investigator, might pose an unacceptable risk by administering study medication
16. The subject received an investigational drug within 30 days prior to inclusion into this study
17. The subject has any current or past medical condition and/or required medication to treat a condition that could affect the evaluation of the study
18. The subject is unwilling or unable to follow the procedures outlined in the protocol
19. The subject is mentally or legally incapacitated

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2014-08; Primary Completion 2015-09 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Effect of linagliptin on vascular inflammation of the carotic artery | up to 6 months
  Examination of the effect of 5 mg linagliptin qd versus placebo on vascular inflammation of the carotic artery by FDG-PET in patients with diabetes mellitus within 6 months.

SECONDARY OUTCOMES:
Effect of linagliptin on vessel wall volume of the carotid artery | baseline and 6 months
  Examination of the effect of 5mg linagliptin qd versus placebo on vessel wall volume of the carotid artery by MRI scan.
Effect of linagliptin on abdominal adipose tissue inflammation | baseline and 6 months
  Evaluation of the effect of 5mg linagliptin qd versus placebo on abdominal adipose tissue inflammation by FDG-PET in addition to adipose tissue biopsies.
Effect of linagliptin on biomarkers of vascular inflammation | baseline and 6 months
  Blood analysis to examine the effect of linagliptin on biomarkers of vascular inflammation.

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaus Marx, Univ.-Prof., Principal Investigator — Department of Internal Medicine I, RWTH Aachen University Hospital
Locations (2):
- Department of Internal Medicine I, University Hospital, Aachen, Germany
- Cardiovascular Research Institute Maastricht (CARIM), Maastricht, Netherlands